CLINICAL TRIAL: NCT07056972
Title: Surveillance Discontinuation in 5 Year Stable Trivial Branch Duct Intraductal Papillary Mucinous Neoplasms (TRIVIAL): International Prospective Single Arm Multicenter Trial
Brief Title: Surveillance Discontinuation in 5 Year Stable Trivial Branch Duct Intraductal Papillary Mucinous Neoplasms
Acronym: TRIVIAL
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Professor, Azienda Ospedaliera di Padova
Other Study IDs: AOP3688
Record Dates: First submitted 2025-06-26; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: IPMN; Pancreatic Cancer
Keywords: ipmn; pancreatic cancer; discontinuation of surveillance
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-arm, discontinuation of follow-up
  Interventions: Other: Discontinuation of surveillance

INTERVENTIONS:
Other: Discontinuation of surveillance — The intervention is discontinuation of current surveillance policies which consist of annual imaging with MRI/MRCP and clinical assessment.

SUMMARY:
BACKGROUND: Patients with trivial branch duct intraductal papillary mucinous neoplasm (BD IPMN) which remain s stable over 5 years reportedly do not have an increased risk of developing pancreatic cancer (PC) compared to the general population. In these patients, d iscontinuation of surveillance seems feasible . However, prospective studies to confirm the safety of this approach are lacking.

AIM: To assess whether current surveillance policies for stable, trivial BD IPMN can be discontinued safely after 5 years of follow up .

METHODS: TRIVIAL is an international prospective multicenter single arm trial exploring discontinuation of surveillance in patients with at least 5 years stable trivial BD IPMN. The trial will include 394 adult patients at least 70 years of age with BD IPMN ≤ 30 millimeter without worrisome features or high risk stigmata during 5 years. The primary endpoint is rate of PC and futile surgery (i.e., surgery for low grade dysplasia IPMN or other non malignant pathology) during 5 year follow up. The predefined target is a rate of 1% and below 3%.

STRENGTHS: The burden for patients to participate in this trial is negligible. P atients will only be asked to answer self reported digital surveys once per year during five years . The potential benefits for patients are twofold: the psychological impact of potentially unnecessary surveillance will be spared to patients , whereas the socio economic burden of repeated imaging will be avoided. Moreover, the study will provide data contributing to the development of new, evidence based surveillance strateg ies At the end of follow up patients undergo MRCP to assess disease course (i.e., development of worrisome features, high risk stigmata, PC).

LIMITATIONS: The most prominent risk of IPMN is the development of pancreatic cancer However this risk will not be omitted fully by the TRIVIAL trial eligibility criteria as participants still have the same risk as the general population. This requires adequate counselling

ELIGIBILITY:
Inclusion Criteria:

* Oral and written informed consent;
* Age ≥70 years;
* BD IPMN with ≥1 dilated branch duct(s) communicating with a nondilated main pancreatic duct (≤5 millimeter) as seen on Magnetic Resonance Cholangio-Pancreatography (MRCP), performed within the last 3 months prior to inclusion;
* At least 5 years of follow up prior to inclusion;
* Absence of relative and absolute indications for surgery at diagnosis and inclusion according to European guidelines;
* Absence of worrisome features and/or high risk stigmata at diagnosis and inclusion according to IAP guidelines;
* Cyst size ≤30 millimeters.

Exclusion Criteria:

* Personal or familial history of pancreatic cancer;
* History of pancreatic surgery;
* Withdrawal of informed consent.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All consecutive patients of ≥70 years of age with trivial BD IPMN ≤30 millimeters that have been stable for at least 5 years are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2031-07-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of pancreatic cancer | Through study completion at 5 years after inclusion
  Primary endpoint is pancreatic cancer (PC), including IPMN derived PC high grade dysplasia (HGD) or concurrent PC, confirmed by pathology (e.g., surgery, fine needle biopsy), at 5 years follow up.
  Concurrent PC is defined as invasive PC that develops independently from the associated IPMN with a non dilated , segment of the pancreatic duct present between the two lesions. Therefore, a clear distinction will be made on what type of PC occurred (i.e., IPMN derived, HGD, concurrent PC).
Incidence of futile surgery | Through study completion at 5 years after inclusion
  Futile surgery is defined as surgery for IPMN with low grade dysplasia (LGD) confirmed at final pathology, or other non malignant diagnosis (i.e., pseudocysts , serous cystadenoma).

SECONDARY OUTCOMES:
Pancreatic cancer related mortality | Through study completion at 5 years after inclusion
All causes mortality | Through study completion at 5 years after inclusion
Time to progression or surgery | Through study completion at 5 years after inclusion
  in months
Incidence of low grade and high grade dysplasia at pathology | Through study completion at 5 years after inclusion
Incidence of individual worrisome and high risk features and of individual relative and absolute indications | Through study completion at 5 years after inclusion
Incidence of pancreatic surgery | Through study completion at 5 years after inclusion
Serum CA 19.9 value | At baseline and through study completion at 5 years after inclusion
  in U/L
Cyst growth | Through study completion at 5 years after inclusion
  mm/year
Adjusted Charlson comorbidity index (ACCI) | At baseline and through study completion at 5 years after inclusion
Rate of misdiagnosis (only in resected patients) patients) | Through study completion at 5 years after inclusion
Incidence of additional follow up and diagnostic work up | Through study completion at 5 years after inclusion
Incidence of symptoms suspect for PC during follow up | Through study completion at 5 years after inclusion